CLINICAL TRIAL: NCT01249638
Title: Randomized, Open, Multicenter Phase III Study With Capecitabine Plus Bevacizumab Versus Capecitabine Plus Irinotecan Plus Bevacizumab as First-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Cap+Bev vs Cap+Iri+Bev 1st-line Therapy in mCRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Volker Heinemann, Prof. Dr. med., University of Munich - Klinikum der Universitaet Muenchen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22011
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2010-11

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Bevacizumab; Capecitabine; Irinotecan; mCRC
MeSH Terms: interventions — Capecitabine; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cap+Bev until PD followed by CAPIRI +Bev (Experimental): Capecitabine + Bevacizumab
  In case of Progression Escalation to:
  Capecitabine + Irinotecan + Bevacizumab
  Interventions: Drug: Capecitabine; Drug: Bevacizumab
- Capiri + Bev (Active Comparator): Capecitabine + Irinotecan + Bevacizumab
  Interventions: Drug: Capecitabine; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine:2 x 1250 mg/m2 day 1-14 followed by 1 week pause q day 21
  Arms: Cap+Bev until PD followed by CAPIRI +Bev
Drug: Bevacizumab — Bevacizumab: 7.5 mg/kg day 1 q day 21
  Arms: Cap+Bev until PD followed by CAPIRI +Bev
Drug: Capecitabine — Capecitabine: 2 x 800mg/m2 day 1-14 followed by 1 week pause q day 21
  Arms: Capiri + Bev
Drug: Irinotecan — Irinotecan: 200 mg/m2 day 1 , q day 21
  Arms: Capiri + Bev
Drug: Bevacizumab — Bevacizumab: 7.5 mg/kg day 1, q day 21
  Arms: Capiri + Bev

SUMMARY:
Patient with multiple metastases, not eligible for surgery, might not profit from intensive chemotherapy regimens. Therefore less intensive regimens focusing on survival and disease control may be a better choice for first line treatment. Therefore this study investigates the combination of capecitabine and bevacizumab versus the combination of capecitabine, bevacizumab and irinotecan. In case of progressive disease, the therapy in patients treated with capecitabine and bevacizumab is intensified by adding irinotecan. Primary endpoint is time-of-failure strategy (TFS) comparing both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum.
* Stage IV disease.
* ECOG 0-1.
* Patients considered suitable for application of chemotherapy.
* Age 18 - 75 years.
* In- or outpatient treatment.
* Estimated life expectancy > 3 months.
* Measurable index lesion according to RECIST criteria. Evaluation of tumor manifestations ≤ 2 weeks prior to treatment start.
* Effective contraception.
* Adequate hematologic function: leukocytes >= 3000/µl, neutrophils >= 1500/µl, platelets >= 100.000/µ, and hemoglobin >= 9g/dl. Bilirubin <= 1,5x upper limit of normal (ULN). ALAT and ASAT <= 2,5x ULN, in case of liver metastases <= 5x ULN. Serum creatinine <= 1,5x ULN.
* No operations within 4 weeks prior to treatment start. No cytologic biopsies within 1 week prior to treatment start. Operation sequels need to be completely healed. Major operations must not be expected at time of study begin, except for potential secondary resection of liver metastases. In case of secondary resection of liver metastases, bevacizumab must be discontinued 6-8 weeks prior to surgery.
* No relevant toxicities due to prior medical treatment at time of study entry.

Exclusion Criteria:

* primary resectable metastases
* heart failure Grade III/IV (NYHA-classification)
* Prior treatment directed against the epidermal growth factor receptor (EGFR).
* Prior treatment with bevacizumab.
* Prior chemotherapy for colorectal cancer, except for adjuvant chemotherapy dating back > 6 months prior to study entry.
* Experimental medical treatment within 30 days prior to study entry.
* Known hypersensitivity reaction to any study medication.
* Pregnant or breast feeding women (pregnancy needs to be excluded by testing of beta-HCG).
* Known or suspected cerebral metastases.
* Clinically significant coronary heart disease, myocardial infarction within the last 12 months or high risk of uncontrolled arrhythmia.
* Acute or subacute ileus, chronic inflammatory bowel disease or chronic diarrhea.
* Abdominal or tracheo-esophageal fistulas, gastrointestinal perforation within 6 months before study entry
* Symptomatic peritoneal carcinosis.
* Severe chronic wounds, ulcera or bone fracture.
* Uncontrolled hypertension.
* Severe proteinuria (nephrotic syndrome).
* Arterial thromboembolic events or hemorrhage within 6 months prior to study entry (except tumor bleeding surgically treated by tumor resection).
* Bleeding diatheses or coagulopathy.
* Full dose anticoagulation.
* Known DPD-deficiency (special screening not required).
* Known glucuronidation-deficiency (special screening not required).
* Contraindication with irinotecan
* Medical history of other malignant disease within 5 years prior to study entry, except for basalioma, and in-situ cervical carcinoma if treated with curative intent.
* Known alcohol or drug abuse.
* Medical or psychiatric condition which contradicts participation of study.
* Limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
TFS | 9 months
  Time of Failure Strategy

SECONDARY OUTCOMES:
ORR, OS, Quality of Life, PFS-1 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Prof. Dr. med., Principal Investigator — University of Munich - Klinikum der Universitaet Muenchen; Sebastian Stintzing, Dr. med., Study Chair — University of Munich - Klinikum der Universitaet Muenchen; Clemens Giessen, Study Chair — University of Munich - Klinikum der Universitaet Muenchen
Locations (1):
- University of Munich - Klinikum der Universitaet Muenchen, Munich, Germany

REFERENCES:
- [Derived] Stahler A, Modest DP, Stintzing S, Borelli B, Keller T, Held S, Fischer von Weikersthal L, Muller L, Graeven U, Decker T, Heintges T, Kahl C, Hoppe B, Kiani A, Kaiser F, Schwaner I, Fruehauf S, Karthaus M, Trarbach T, Klauschen F, Horst D, Cremolini C, Heinemann V. Individual Patient Data Meta-Analysis of Consensus Molecular Subtypes as Biomarkers of First-Line Treatment in RAS Wild-Type Metastatic Colorectal Cancer. J Clin Oncol. 2026 Jan;44(1):31-41. doi: 10.1200/JCO-25-00596. Epub 2025 Nov 18. PMID 41252656
- [Derived] Stahler A, Modest DP, Fischer von Weikersthal L, Kaiser F, Decker T, Held S, Graeven U, Schwaner I, Denzlinger C, Schenk M, Kurreck A, Heinrich K, Giessen-Jung C, Neumann J, Kirchner T, Jung A, Stintzing S, Heinemann V. First-line fluoropyrimidine plus bevacizumab followed by irinotecan-escalation versus initial fluoropyrimidine, irinotecan and bevacizumab in patients with metastatic colorectal cancer - Final survival and per-protocol analysis of the randomised XELAVIRI trial (AIO KRK 0110). Eur J Cancer. 2022 Sep;173:194-203. doi: 10.1016/j.ejca.2022.06.019. Epub 2022 Aug 5. PMID 35940054
- [Derived] Stahler A, Heinemann V, Schuster V, Heinrich K, Kurreck A, Giessen-Jung C, Fischer von Weikersthal L, Kaiser F, Decker T, Held S, Graeven U, Schwaner I, Denzlinger C, Schenk M, Neumann J, Kirchner T, Jung A, Kumbrink J, Stintzing S, Modest DP. Consensus molecular subtypes in metastatic colorectal cancer treated with sequential versus combined fluoropyrimidine, bevacizumab and irinotecan (XELAVIRI trial). Eur J Cancer. 2021 Nov;157:71-80. doi: 10.1016/j.ejca.2021.08.017. Epub 2021 Sep 8. PMID 34507244
- [Derived] Heinrich K, Modest DP, Ricard I, Fischer von Weikersthal L, Decker T, Kaiser F, Graeven U, Uhlig J, Schenk M, Freiberg-Richter J, Peuser B, Denzlinger C, Giessen-Jung C, Stahler A, Michl M, Held S, Jung A, Kirchner T, Stintzing S, Heinemann V. Gender-dependent survival benefit from first-line irinotecan in metastatic colorectal cancer. Subgroup analysis of a phase III trial (XELAVIRI-study, AIO-KRK-0110). Eur J Cancer. 2021 Apr;147:128-139. doi: 10.1016/j.ejca.2021.01.025. Epub 2021 Feb 27. PMID 33647548
- [Derived] Modest DP, Fischer von Weikersthal L, Decker T, Vehling-Kaiser U, Uhlig J, Schenk M, Freiberg-Richter J, Peuser B, Denzlinger C, Peveling Genannt Reddemann C, Graeven U, Schuch G, Schwaner I, Stahler A, Jung A, Kirchner T, Held S, Stintzing S, Giessen-Jung C, Heinemann V; XELAVIRI/AIO KRK0110 Investigators. Sequential Versus Combination Therapy of Metastatic Colorectal Cancer Using Fluoropyrimidines, Irinotecan, and Bevacizumab: A Randomized, Controlled Study-XELAVIRI (AIO KRK0110). J Clin Oncol. 2019 Jan 1;37(1):22-32. doi: 10.1200/JCO.18.00052. Epub 2018 Nov 2. PMID 30388045
- [Derived] Giessen C, von Weikersthal LF, Hinke A, Stintzing S, Kullmann F, Vehling-Kaiser U, Mayerle J, Bangerter M, Denzlinger C, Sieber M, Teschendorf C, Freiberg-Richter J, Schulz C, Modest DP, Moosmann N, Aubele P, Heinemann V. A randomized, phase III trial of capecitabine plus bevacizumab (Cape-Bev) versus capecitabine plus irinotecan plus bevacizumab (CAPIRI-Bev) in first-line treatment of metastatic colorectal cancer: the AIO KRK 0110 trial/ML22011 trial. BMC Cancer. 2011 Aug 23;11:367. doi: 10.1186/1471-2407-11-367. PMID 21861888